CLINICAL TRIAL: NCT06831916
Title: Effects of Hemp-Derived Cannabinoids on Menopause Symptoms
Brief Title: Impact of Cannabinoids on Menopause Symptoms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Terra Mater Botanicals Pty Ltd (Unknown)
Responsible Party: Principal Investigator, Carrie Cuttler, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20779-001
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Perimenopause; Menopause
Keywords: Menopause; Perimenopause; Cannabinoids; CBG; CBD; Cognition; Anxiety; Sleep; Pain; Mood; Stress; Brain Fog
MeSH Terms: conditions — Anxiety Disorders; Pain; Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistants who administer the protocol will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Participants in this arm will receive a placebo.
  Interventions: Other: Placebo
- Active Arm (Experimental): Participants in this arm will receive an active product.
  Interventions: Dietary Supplement: Active Cannabinoid Product

INTERVENTIONS:
Dietary Supplement: Active Cannabinoid Product — Participants will be administered a product with minor cannabinoids and terpenes.
  Arms: Active Arm
Other: Placebo — Participants will be administered a placebo.
  Arms: Placebo Arm

SUMMARY:
The purpose of the study is to examine the impact of the hemp-derived minor cannabinoids on symptoms of menopause/perimenopause.

DETAILED DESCRIPTION:
This study implements a randomized, double-blind, placebo-controlled, observational field experiment design to examine the impact of hemp-derived minor cannabinoids on symptoms of menopause/perimenopause. The study will require 3 months to complete.

Healthy adult women (between the ages of 40-60) experiencing psychological and physical symptoms of menopause or perimenopause will be recruited via advertisements on social media, physicians' offices, in the community, at menopause conferences/conventions, and on internet forums. Prospective participants will complete a brief online screening survey to determine whether they meet eligibility requirements. Eligible participants will be asked to provide their first name and phone number if they want to be contacted via text message to participate.

Initial Zoom Session: Eligible participants who agree to participate will be asked to schedule an initial Zoom session, during which they will provide informed consent, review the study requirements, and complete cognitive tests including tests of memory and verbal fluency. Tests include the Rey Auditory Verbal Learning Test (RAVLT), FAS Verbal Fluency Test, Digit Span Forward and Backward (DSF, DSB), Deese-Roediger-McDermott Paradigm (DRM), Corsi Forward and Backward, and Prospective Memory (PM) Tasks. They will also be given the contact information for a company that manufactures and distributes hemp-derived cannabinoids. Participants will be asked to contact the company and request that they directly ship the product to them (the participant). The product will be provided at no cost to the participant (or to the PI or their lab). The PI will randomize each participant to the active or placebo condition and will subsequently contact the distributor to inform them of which product to ship (active or placebo). Participants will be given a link to an online Qualtrics survey that will be used to assess demographic characteristics, medications, and menopause/perimenopause symptoms, including depression, anxiety, perceived stress, physical and emotional health, insomnia, and everyday memory problems (Beck Depression Inventory [BDI], Beck Anxiety Inventory [BAI], Perceived Stress Scale [PSS], Short Form Health Survey [SF-36], Insomnia Severity Index [ISI], and Everyday Memory Questionnaire [EMQ], respectively).

Baseline: Participants will then complete four weeks of baseline assessments via ecological momentary assessment (EMA). Specifically, twice a day: shortly after they eat breakfast, and shortly after they eat dinner participants will complete a brief survey on their phone. For each EMA survey, they will be asked to indicate whether they experienced various emotional/psychological symptoms of menopause as well as whether they experienced various physical symptoms of menopause since their last EMA assessment. For each endorsed symptom, they will be asked to rate its severity as well as how much it interfered with their life using a 0 to 10 visual analog scale. In the morning survey, they will also be asked to indicate how well they slept the night before. Once a week, participants will also complete a series of EMA cognitive tests, including tests of verbal memory, spatial memory, working memory, inhibition, psychomotor speed, and attention (assessed using NeuroUX's Memory List, CopyKat, 2-Back, Digit Symbol Substitution, Color Names, Quick Tap Level 1and 2, and Trail Making A and B). Participants will be sent text messages with a link to the tests and will be instructed to complete them on their smartphone. At the end of the month, participants will meet a researcher over Zoom where they will complete additional cognitive tests (RAVLT, FAS, DSF/DSB, DRM, Corsi, PM). Cognitive tests involving word lists or letter sets (i.e., RAVLT, FAS, DRM) will be counterbalanced using a Latin Square design. At the end of the session, they will be sent a link to complete an online survey that will be used to assess menopause/perimenopause symptoms, including depression, anxiety, perceived stress, physical and emotional health, insomnia, and everyday memory problems (BDI, BAI, PSS, SF-36, ISI, EMQ, respectively). This period of time constitutes the baseline assessment period.

Phase 1: Phase 1 will begin after 4 weeks of baseline assessments and will continue for 4 weeks. During this phase, participants will be asked to take a single dose of the active or placebo version of the product (in a double-blind manner) twice a day (once after breakfast and again after dinner) and to complete EMA survey assessments twice a day (after orally ingesting each dose). Participants will be sent reminders and links via text message. For each EMA survey, they will be asked to indicate whether they took the study product, and if so what time they took the product. If they indicate they have not taken the product yet they will instructed to do so or provide a reason why they cannot do so. Next, they will be asked to indicate whether they experienced various emotional symptoms of menopause/perimenopause as well as whether they experienced various physical symptoms of menopause/perimenopause since their last EMA survey assessment. For each endorsed symptom, they will be asked to rate its severity as well as how much it interfered with their life using a 0 to 10 visual analog scale. In the morning survey, they will also be asked to indicate how well they slept the night before. Participants will also report on whether they experienced any side effects. Once a week, participants will also complete a series of EMA cognitive tests, including tests of verbal memory, spatial memory, inhibition, psychomotor speed, and attention (assessed using NeuroUX's Memory List, CopyKat, 2-Back, Digit Symbol Substitution, Color Names, Quick Tap Level 1and 2, and Trail Making A and B). Participants will be sent text messages with a link to the tests and will be instructed to complete them on their smartphone. At the end of the four weeks, participants will meet a researcher over Zoom where they will complete additional cognitive tests (RAVLT, FAS, DSF/DSB, DRM, Corsi, PM). They will also be asked if they would like to double the dose of the tincture for Phase 2 and additional product will be sent to participants who indicate they want to increase the dose. At the end of the session, they will be sent a link to complete an online survey that will be used to assess menopause/perimenopause symptoms, including depression, anxiety, perceived stress, physical and emotional health, insomnia, and everyday memory problems (BDI, BAI, PSS, SF-36, ISI, EMQ, respectively).

Phase 2: Phase 2 will begin after 4 weeks of phase 1 assessments and will continue for 4 weeks. During this phase, participants will be asked to take two doses of the active or placebo version of the product (in a double-blind manner) twice a day (once after breakfast and again after dinner) if they indicated they wanted to increase the dose of the product. Otherwise, they will continue taking a single dose twice a day. They will complete the same EMA survey assessments twice a day (after orally ingesting each dose). Participants will be sent reminders and links via text message. For each EMA survey they will be asked to indicate whether they took the study product, and if so what time they took the product. If they indicate they have not taken the product yet they will instructed to do so or provide a reason why they cannot do so. Next, they will be asked to indicate whether they experienced various emotional symptoms of menopause/perimenopause as well as whether they experienced various physical symptoms of menopause/perimenopause since their last EMA survey assessment. For each endorsed symptom, they will be asked to rate its severity as well as how much it interfered with their life using a 0 to 10 visual analog scale. In the morning survey, they will also be asked to indicate how well they slept the night before. Participants will also report on whether they experienced any side effects. Once a week, participants will also complete a series of cognitive tests using EMA, including tests of verbal memory, spatial memory, inhibition, psychomotor speed, and attention (assessed using NeuroUX's Memory List, CopyKat, 2-Back, Digit Symbol Substitution, Color Names, Quick Tap Level 1and 2, and Trail Making A and B). Participants will be sent text messages with a link to the tests and will be instructed to complete them on their smartphone. At the end of the four weeks, participants will meet a researcher over Zoom where they will complete additional cognitive tests (RAVLT, FAS, DSF/DSB, DRM, Corsi, PM). At the end of the session, they will be sent a link to complete the online survey (including the BDI, BAI, PSS, SF-36, ISI, and EMQ). The study ends after phase 2.

ELIGIBILITY:
Inclusion Criteria:

* designated female at birth
* 40-60 years of age
* able to give informed consent (no intellectual disability)
* stable pharmacotherapeutic regimen, no change in the past 3 months
* abstinent from regular cannabis use (<1x/month) for past year, and willing to abstain from use for 3 months
* abstinent for supplements, don't add any supplements (no changes in past 3 months)
* own a smartphone
* have access to Zoom on a secure, stable internet connection
* perimenopausal or menopausal

Exclusion Criteria:

* currently taking anti-depressant, anti-anxiety, and/or antipsychotic medication
* severe depression, neurovegetative symptoms, or current suicidality
* psychosis or family history of psychosis
* pregnant or breastfeeding
* chemotherapy
* hypotension
* drug testing for work or other reasons
* illicit drug use in past 3 months (cannabis not illicit)
* heavy alcohol use (4 drinks more than 4x/week)
* international/air travel planned for more than one week in the next 3 months

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Depression Monthly Assessment: Beck Depression Inventory | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the Beck Depression Inventory (BDI). Participants will complete the BDI after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Anxiety Monthly Assessment: Beck Anxiety Inventory | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the Beck Anxiety Inventory (BAI). Participants will complete the BAI after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Perimenopausal Depression Monthly Assessment: Meno-D | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the Meno-D. Participants will complete the Meno-D after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Emotional/Mental Symptoms Daily Assessment | Emotional/mental symptoms will be assessed during each session (morning and night) of the daily EMA assessments, for the 3 month duration of the study.
  During each EMA session (twice daily), participants will be asked to indicate emotional/mental symptoms they have experienced since the last time they completed the survey. Possible symptoms include: new or worsening anxiety; new or worsening depression/crying; loss of interest in most things; fatigue or loss of energy; diminished self-esteem; mood swings; irritability; brain fog. They will also have the opportunity to write in other symptoms experienced.
  For each endorsed symptom, participants will be asked to rate the severity (on a 0 to 10 visual analog scale) and the degree to which that symptom interferes with their life (on a 0 to 10 visual analog scale).

SECONDARY OUTCOMES:
Physical Symptoms Daily Assessment | Physical symptoms will be assessed during each session (morning and night) of the daily EMA assessments, for the 3 month duration of the study.
  During each EMA session (twice daily), participants will be asked to indicate physical symptoms they have experienced since the last time they completed the survey. Possible symptoms include: hot flushes/flashes or night sweats; headaches/migraines; feeling dizzy or faint; muscle or joint pain or weakness; breast tenderness or pain; heart palpitations or a racing heart; vaginal dryness or pain; urinary frequency, urgency, leaking, and/or urinary tract infections. They will also have the opportunity to write in other symptoms experienced.
  For each endorsed symptom, participants will be asked to rate the severity (on a 0 to 10 visual analog scale) and the degree to which that symptom interferes with their life (on a 0 to 10 visual analog scale).
  High-risk responses (i.e., severe symptoms) will alert the PI and relevant resources/information will be provided.
Side Effects Daily Assessment | Side effects will be assessed during each session (morning and night) of the daily EMA assessments, for the 3 month duration of the study.
  During each EMA session (twice daily), participants will be asked to indicate any side effects they have experienced since the last time they completed the survey. Possible side effects include: dry eyes; dry mouth; dizziness, sleepiness or fatigue, increased appetite, racing heart or heart palpitations, anxiety, feeling intoxicated; feeling impaired; and difficulty urinating.
Verbal Memory Monthly Assessment: RAVLT | The RAVLT will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  Participants will complete the Rey Auditory Verbal Learning Test (RAVLT) at each monthly assessment. The RAVLT will be administered via Zoom by a research assistant at the beginning of the study, after four weeks of a baseline phase, and at the end of both phase 1 and phase 2. Four alternate versions will be administered in a counterbalanced manner.
Verbal Fluency Monthly Assessment: FAS | The FAS verbal fluency test will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  Participants will complete a verbal fluency assessment at each monthly assessment. The FAS verbal fluency test will be administered via Zoom by a research assistant at the beginning of the study, after four weeks of a baseline phase, and at the end of both phase 1 and phase 2. Four alternate letter sets will be administered in a counterbalanced manner.
ST/Working Memory Monthly Assessment: Digit Span Forward and Backwards | The digit span tests will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  Participants will complete the digit span forward and backward tests at each monthly assessment. The test will be administered via Zoom by a research assistant at the beginning of the study, after four weeks of a baseline phase, and at the end of both phase 1 and phase 2.
False Memory Monthly Assessment: Deese-Roediger-McDermott Paradigm | The false memory test will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  Participants will complete the Deese-Roediger-McDermott Paradigm false memory test at each monthly assessment. The test will be administered via Zoom by a research assistant at the beginning of the study, after four weeks of a baseline phase, and at the end of both phase 1 and phase 2. Four alternate versions will be administered in a counterbalanced manner.
ST/Working Spatial Memory Monthly Assessment: Corsi Forward and Backward | The Corsi tests will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  Participants will complete the Corsi block-tapping tests (forward and backward) at each monthly assessment. The test will be administered via Zoom by a research assistant at the beginning of the study, after four weeks of a baseline phase, and at the end of both phase 1 and phase 2.
Prospective Memory Monthly Assessment: Difficulty Ratings | The prospective memory tests will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At each monthly Zoom session, participants will be asked to try to remember to rate the difficulty of each cognitive test completed during the session immediately after completing each test. Instructions and a 0 through 10 visual analog scale will be provided at the beginning of the session. Participants will not be reminded to provide ratings.
Prospective Memory Monthly Assessment: Survey Completion | The prospective memory tests will be administered during monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link and will be asked to email the RA once they have completed the survey. Instructions and the RA's email address will be provided immediately before sending the survey link and logging off of Zoom. Participants will not be reminded to email the RA.
Brain Fog Monthly Assessment: Everyday Memory Questionnaire | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the Everyday Memory Questionnaire (EMQ). Participants will complete the EMQ after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Stress Monthly Assessment: Perceived Stress Scale | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the Perceived Stress Scale (PSS). Participants will complete the PSS after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Health Monthly Assessment: SF-36 Health Survey Questionnaire | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the SF-36 Health Survey Questionnaire. Participants will complete the SF-36 after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Sleep Monthly Assessment: Insomnia Severity Index | The survey will be completed shortly after the monthly Zoom sessions, during four different sessions. They will occur at approximately week 1, 5, 9, and 13.
  At the end of each monthly Zoom session, participants will be sent a survey link including the Insomnia Severity Index (ISI). Participants will complete the ISI after each zoom session, including the first session, the baseline session after four week, and after both phase 1 and phase 2.
Sleep Daily Assessment | Sleep quality will be assessed during each morning session of the daily EMA assessments, for the 3 month duration of the study.
  During each morning EMA session, participants will be asked to rate how well they slept the previous night on a 0 to 10 visual analog scale.
Verbal Memory Weekly Assessment: Memory List | Verbal memory will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "Memory List" game, assessing verbal memory. The total cognitive assessment is designed to take around 15 minutes.
Spatial Memory Weekly Assessment: CopyKat | Spatial memory will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "CopyKat" game, assessing spatial memory. The total cognitive assessment is designed to take around 15 minutes.
Working Memory Weekly Assessment: 2-Back | Working memory will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "2-Back" game, assessing working memory. The total cognitive assessment is designed to take around 15 minutes.
Digit Symbol Substitution Weekly Assessment: Digit Symbol Task | Digit symbol substitution ability will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "Digit Symbol Task" game, assessing processing speed, and attention. The total cognitive assessment is designed to take around 15 minutes.
Simple Reaction Time Weekly Assessment: Quick Tap Level 1 | Simple reaction time will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "Quick Tap Level 1" game, assessing simple reaction time. The total cognitive assessment is designed to take around 15 minutes.
Working Memory/Attention Weekly Assessment: Color Names | "Color Names" performance will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "Color Names" game (i.e., Stroop test) assessing executive functioning (inhibitory control). The total cognitive assessment is designed to take around 15 minutes.
Trail Making Test Weekly Assessment: A and B | Trail making ability will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "Trail Making A" game (letter sequencing) and "Trail Making " game (letter-number alternating sequencing) assessing attention and cognitive flexibility (B). The total cognitive assessment is designed to take around 15 minutes.
Response Inhibition Weekly Assessment: Quick Tap Level 2 | Response inhibition will be assessed during the weekly EMA cognitive assessments. Participants will be prompted to complete these games during their morning daily EMA session, for the 3 month duration of the study.
  During the weekly EMA cognitive assessments, participants will complete NeuroUX's "Quick Tap Level 2" game (i.e., Go-No-Go), inhibitory control. The total cognitive assessment is designed to take around 15 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University - Pullman Campus, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request and after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will be retained indefinitely.
Access Criteria: Researchers wanting to conduct secondary data analysis following my own publication.